CLINICAL TRIAL: NCT06801587
Title: Preemptive Co-infiltration of Triamcinolone Acetonide With Ropivacaine for Postoperative Pain in Patients Undergoing Major Spinal Surgery
Brief Title: Preemptive Co-infiltration of Triamcinolone Acetonide With Ropivacaine for Postoperative Pain in Major Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fang Luo (Other)
Responsible Party: Sponsor-Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY-2019-112-02-4
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pain; Postoperative
MeSH Terms: conditions — Pain | interventions — Triamcinolone Acetonide; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triamcinolone acetonide plus ropivacaine group (Experimental): The local infiltration solution in the triamcinolone acetonide plus ropivacaine group will consist of triamcinolone acetonide and ropivacaine.
  Interventions: Drug: Triamcinolone acetonide plus ropivacaine
- The ropivacaine alone group (Active Comparator): The local infiltration solution in the ropivacaine alone group will consist of ropivacaine alone.
  Interventions: Drug: Ropivacaine alone

INTERVENTIONS:
Drug: Triamcinolone acetonide plus ropivacaine — The local infiltration solution in the triamcinolone acetonide plus ropivacaine group will consist of ropivacaine and triamcinolone acetonide. For local infiltration, a total of 30mL solution will be prepared for each group, 1 ml of triamcinolone acetonide (40mg per 1ml) plus 15 ml of 1% ropivacaine diluted to 30 ml with saline as the test drug in the triamcinolone acetonide group. The surgeon will perform incision infiltration before the skin incision. A total of 10 mL of solution will be injected into each level. The study solution will be injected into the entire thickness of the planned incision site. The epidural space and intrathecal space will not be infiltrated.
  Arms: Triamcinolone acetonide plus ropivacaine group
Drug: Ropivacaine alone — The local infiltration solution in the ropivacaine alone group will consist of ropivacaine alone. For local infiltration, a total of 30mL solution will be prepared for each group, which will include 15ml of ropivacaine added to 15mL of saline for ropivacaine group . The surgeon will perform incision infiltration before the skin incision. A total of 10 mL of solution will be injected into each level. The study solution will be injected into the entire thickness of the planned incision site. The epidural space and intrathecal space will not be infiltrated.
  Arms: The ropivacaine alone group

SUMMARY:
Patients undergoing major spinal surgery usually experience moderate to-severe postoperative pain. Inadequate pain control may lead to severe complications.

Local infiltration analgesia (LIA) with a local anesthetic, is a simple, minimally invasive, and effective postoperative pain management technique. However, LIA with local anesthetic alone can only last for a short time, steroid as adjuvant can enhance postoperative analgesia and prolong postoperative analgesia time. Triamcinolone acetonide as an adjunctive infiltration to local anesthesia presented a superior analgesic benefit compared with local anesthesia alone in various types of surgeries. To date, no studies have evaluated the additive analgesia effects of triamcinolone acetonide on incision infiltration in major spinal surgery. The purpose of this trial is to determine whether preemptive co-infiltration of triamcinolone acetonide and ropivacaine in surgical incision will further reduce postoperative opioid requirements and pain score after spinal surgery than that of ropivacaine alone.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years; Patients scheduled for elective laminoplasty or laminectomy with no more than 3 levels under general anesthesia; American Society of Anesthesiologists (ASA) physical status of I-III; Anticipated full recovery and cooperation within 2 hours postoperatively.

Exclusion Criteria:

History of spinal surgery; Inability to use a patient-controlled analgesia (PCA) pump or comprehend the pain visual analog scale (VAS); Body mass index (BMI)<15kg/m2 or >35kg/m2; Peri-incisional infection; History of diabetes mellitus and other metabolic diseases; History of severe cardiopulmonary, hepatic or renal dysfunction; Preoperative coagulation abnormalities (activated partial thromboplastin time greater than 1.5 times normal value); History of allergies to any of the study drugs; History of alcohol or drugs abuse (more than 2 weeks), or use of any analgesic within 24h before surgery; Use of systemic steroids within 1 week before surgery; History of psychiatric disorders, chronic neck or back pain; History of radiation therapy and chemotherapy or with a high probability of such treatment postoperatively; Pregnant or breastfeeding; Refusal to sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
The cumulative consumption of sufentanil within 24 hours after spinal surgery via the PCA pump. | Within 24 hours after spinal surgery
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) pump. Participates will be advised to push the analgesic demand button if they feel pain

SECONDARY OUTCOMES:
The cumulative consumption of sufentanil via PCA pump between 24 hours and 48 hours postoperatively. | Between 24 hours and 48 hours after spinal surgery
  Patients will use PCA device for pain management within the the first 48 hours after surgery. When the patients feel pain, the PCA button will be pressed. When the patients feel no pain, the PCA button will not be pressed. The PCA pump will provide a bolus of 2μg sufentanil with a 10 minutes lock-out time, and the maximum dose of sufentanil will be limited to 8μg/h.
Number of patients without PCA press button | Within 48 hours after spinal surgery
  Patients will use PCA device for postoperative analgesia. When the patients feel pain, the PCA button will be pressed. When the patients feel no pain, the PCA button will not be pressed. The PCA pump will provide a bolus of 2μg sufentanil with a 10 minutes lock-out time, and the maximum dose of sufentanil will be limited to 8μg/h.
The time of first PCA demand | Within 48 hours after spinal surgery
  The first time that the participants press PCA button.
The total number of PCA presses including both valid and invalid presses | Within 48 hours after spinal surgery
  The total number that participants press PCA button including valid and invalid presses
Postoperative visual analogue scale (VAS) score during movement(VASm) | At 2 hours, 4 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 3 weeks, 1 month and 3 months postoperatively
  The pain will be assessed by VAS scores during movement (0 indicates no pain, 10 indicates the most severe pain imaginable, a higher score means worse pain)
Postoperative VAS score at rest(VASr) | At 2 hours, 4 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 3 weeks, 1 month and 3 months postoperatively
  The pain will be assessed by VAS scores at rest (0 indicates no pain, 10 indicates the most severe pain imaginable, a higher score means worse pain)
Total consumption of Tylenol as supplementary analgesia | Four separate postoperative periods ( 0- postoperative 48 hours, postoperative 48 hours-postoperative 2 weeks, postoperative 2 weeks-postoperative 1 month, and postoperative 1 month-postoperative 3 months)
  During the initial postoperative 48 hours, when VAS>4 (either VASm or VASr) after pressing button four times with PCA pump for pain relief, patients will be treated for supplementary analgesia with oral Tylenol (Mallinckrodt Inc.), a combination of 5mg of oxycodone hydrochloride and 325mg paracetamol per tablet at a minimum interval of 6 hours. After the initial postoperative 48 hours, patients will be allowed to take oral Tylenol as needed (dose as previously described), until the end of the study (3-months follow-up).
Patient Satisfaction Score (PSS) with pain relief | At 48 hours, 72 hours, 1 week, 2 weeks, 3 weeks 1 month and 3 months postoperatively
  4 scales; never, sometimes, usually or always
Postoperative nausea and vomiting (PONV) score | At 2 hours, 4 hours, 24 hours, 48 hours and 72 hours postoperatively
  The Postoperative Nausea and Vomiting (PONV) will be measured using an ordinal scale, with 0 indicating no nausea; 1, mild nausea not requiring treatment; 2, nausea requiring treatment; 3, vomiting.
Ramsay Sedation Scale (RSS) | At 2 hours, 4 hours, 24 hours, 48 hours and 72 hours postoperatively
  The Ramsay Sedation Scale (RSS): A 6-point scale will be used to assess sedation levels, with 1 indicating agitated, anxious; 2, cooperative; 3, only responds to commands; 4, strong response to glabellar tapping or noisy stimulants; 5, weak response to glabellar tapping or noisy stimulants; 6, no response.
Patient Scar Assessment and the Observer Scar Assessment Scale (POSAS) | At 2 weeks, 1 month and 3 months postoperatively
  The POSAS consists of an Observer and a Patient Scale and includes a comprehensive list of items, based on clinically relevant scar characteristics. The observer scores six items: vascularization, pigmentation, thickness, surface roughness, pliability, and surface area. The patient scores six items: pain, pruritus, color, thickness, relief, and pliability. All included items are scored on the same polytomous 10-point scale, in which a score of 1 is given when the scar characteristic is comparable to normal skin and a score of 10 reflects the worst imaginable scar. All items are summed to give a total scar score, and therefore, a higher score represents a poorer scar quality.
Rate of steroid-related side effects and complications | Through the whole follow-up, an average of 3 months
  Steroid-related side effects (hyperglycemia, gastrointestinal bleeding, gastritis, etc.) or complications including any cardiac, respiratory, renal, neurologic, or infection complications occured during the hospitalization.
Readmission rate within 3 months after spine surgery | Through the whole follow-up, within 3 months after spine surgery
  Patients readmitted within 3 months after spine surgery
Length of Postoperative Anesthesia Care Unit (PACU) stay | Approximately 30 minutes to 2 hours after surgery
  Time from arrival at PACU after tracheal extubation to transfer from PACU to the surgical ward (modified Aldrete score ≥9).
Duration of hospitalization after surgery | Approximately 1-2 weeks after surgery
  Duration of hospitalization after surgery (time required from the end of surgery to discharge from the hospital).
Total consumption of remifentanil during surgery | During surgery
  Total remifentanil dosages during surgery
Total consumption of loxoprofen | From postoperative 48 hours to approximately 1-2 weeks after surgery
  Pain management will be provided via the sufentanil PCA device for the first 48 hours following surgery. After that, patients will switch to taking oral loxoprofen 60 mg at a minimum interval of 8 hours and a maximum 180mg per day as needed until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol